CLINICAL TRIAL: NCT00453596
Title: Analysis of Implantation Failure and Establishment of Therapy for Implantation Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yamaguchi University Hospital (Other)
Other Study IDs: 16520
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2007-03-29 (Estimated); Status verified 2007-03

CONDITIONS: Infertility
Keywords: infertile women; thin endometrial thickness; implantation failure
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Impaired endometrial growth (thin endometrial thickness) is a critical factor for implantation failure. In this study, effects of vitamin E on endometrial growth are studied.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial thickness < 8 mm

Exclusion Criteria:

* Women with fibroids
* Women receiving hormone therapy

Sex: Female
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Norihiro Sugino, M.D., PhD., Study Chair — Yamaguchi University Hospital
Locations (1):
- Yamaguchi University Hospital, Ube, Japan